CLINICAL TRIAL: NCT05929976
Title: Multi-National Nutritional Biobanking Program in Pediatric Oncology InterNatIonal CHildhood Leukemia Microbiome/MEtabolome Cohort
Brief Title: InterNatIonal CHildhood Leukemia Microbiome/MEtabolome Cohort
Acronym: NICHE
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: International Agency for Research on Cancer (Other)
Responsible Party: Principal Investigator, Elena Ladas, Professor, Columbia University
Other Study IDs: AAAU1407
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia; Nutrition Aspect of Cancer; Microtia; Genetic Predisposition
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Microtia; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood will be collected at diagnosis, end of induction, beginning of maintenance, end of treatment, and 1 year post end of treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Nutritional status is a measurable and modifiable factor that is often not considered during treatment and its clinical impact undervalued due in part to the heavy demands on clinicians in low and middle income countries to deliver therapy to large numbers of patients. The proposed study will create a biobank of clinical data and biological specimens which will foster future studies on cancer progression and prognosis as well as toxicities during treatment which may impact survivorship and late-effects. Eligible patients must be between 3 years and 18 years of age at time of assent/consent, have newly diagnosed B- or T-cell acute lymphoblastic leukemia or mixed phenotype acute leukemia confirmed by pathology report, and must be receiving treatment at one of the participating centers. Patients receiving hematopoietic cell transplant will be excluded. Institutions were selected to ensure representation of several global health indicators related to nutritional status and wealth classification according to the World Bank. Data related to demographic variables (socioeconomic status, food security), lifestyle habits (diet, physical activity), nutritional anthropometrics (height, weight and arm anthropometry), and nutritional biological indices (stool and blood) will be collected at designated timepoints throughout treatment and one year after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 3 years and 18 years of age at time of assent/consent.
* Patients must have newly diagnosed B- or T-cell ALL, or mixed phenotype acute leukemia confirmed by pathology report.
* Patients must be receiving treatment at one of the participating centers.

Exclusion Criteria:

- Patients receiving hematopoietic cell transplant.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents diagnosed with acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 4900 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Create a prospective multinational biorepository of pediatric specimens (stool, blood) obtained at diagnosis, end of induction, beginning of maintenance, end of treatment, and 1-year after treatment among children/adolescents with ALL. | 7 years
Collect sociodemographic data at sequential timepoints during treatment for ALL. | 7 years
Collect dietary data at sequential timepoints during treatment for ALL. | 7 years
Collect physical activity data at sequential timepoints during treatment for ALL. | 7 years
Collect clinical information (disease characteristics, treatment-related toxicities, survival) at sequential timepoints during treatment for ALL to accompany the biorepository of blood and stool specimens. | 7 years
Collect nutritional anthropometrics at sequential timepoints during treatment for ALL to accompany the biorepository of blood and stool specimens. | 7 years

CONTACTS AND LOCATIONS:
Locations (8):
- Columbia University Irving Medical Center, New York, New York, United States
- Brazil (3):
  - Hospital de Cancer Infanto Juvenil de Barretos, Barretos
  - Instituto de Medicina Integral Prof. Fernando Figueira (IMIP), Recife
  - Instituto de Tratamento do Câncer Infantil (ITACI), São Paulo
- Unidad Nacional De Oncologia Pediatrica, Guatemala City, Guatemala
- Hospital Escuela, Tegucigalpa, Honduras
- Post-Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India
- Muhumbili Hospital, Dar es Salaam, Dar es Salaam Region, Tanzania

IPD SHARING:
Plan to Share IPD: No